CLINICAL TRIAL: NCT00281034
Title: Outcome Assessment Using SF-36 v2 in Stroke Patient Study(OASIS Study)
Brief Title: OASIS STUDY Outcome Assessment Using SF-36 v2 in Stroke Patient Study(OASIS STUDY)
Status: Completed | Type: Observational
Sponsor: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Yukito Shinohara, Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Kyorin Pharmaceutical Co.,Ltd
Other Study IDs: OASIS-2005; oasis-2007
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Stroke
Keywords: brain infarction; SF-36; HRQOL; Japan; Post-stroke syndrome
MeSH Terms: conditions — Stroke; Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OASIS Study Group

SUMMARY:
1. To survey the health-related quality of life using the SF-36v2 score of patients with chronic brain infarction in Japan
2. Chronic brain infarction in Japan is better than EU/USA

DETAILED DESCRIPTION:
Period:2005-2007

Observation Time:baseline, 8week, 24week

matters investigated:

1. QOL determination using SF-36 v2
2. Age, sex, brain infarction type, stroke severity (modified Rankin scale), side of stroke, complication, smoking, alcohol, dizziness-vertigo-presyncope-light headedness, combination medicine, subjective symptoms, psychic symptoms, rehabilitation, recurrence, evaluation of depression (Japan-Stroke Scale (JSS)-D)

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose last attack occurred more than 1 month ago
2. Outpatients (including hospitalization for rehabilitation)
3. Japanese nationality
4. Patients who consented to participate in this study
5. Group I: Patients with dizziness, vertigo, presyncope, and light-headedness which are likely due to secondary chronic cerebral circulation impairment associated with sequelae of brain infarction, and patients for whom KETAS (IBUDILAST) was prescribed Group II: Patients without dizziness, vertigo, presyncope, and light-headedness which are likely due to chronic cerebral circulation impairment associated with sequelae of brain infarction

Exclusion Criteria:

1. Patients who cannot read, understand and fill in the questionnaire by themselves
2. Patients who idle their time away
3. Patients who are hospitalized
4. Patients who are undergoing treatment for dizziness, vertigo, presyncope, light-headedness which are likely due to chronic cerebral circulation impairment associated with sequelae of brain infarction
5. Patients whose dizziness, vertigo, presyncope, and light-headedness is definitely or likely caused by Meniere disease, vestibular neuronitis, benign paroxysmal positional vertigo, otitis media, or epilepsy6. Patients whom the investigator judges are not suitable to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Univercity, Main hospital, general Hospital,0pen
Sampling Method: Probability Sample
Enrollment: 2069 (Actual)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
score of SF-36 | 0, 8 week, 24 week

CONTACTS AND LOCATIONS:
Overall Officials: Yukito Shinohara, MD, Study Chair — Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital
Locations (1):
- Federation of National Public Service Personnel Mutual Aid Associations Tachikawa Hospital, Tachikawa, Tokyo, Japan

REFERENCES:
- [Derived] Shinohara Y; OASIS Study Group. Factors affecting health-related quality of life assessed with the SF-36v2 health survey in outpatients with chronic-stage ischemic stroke in Japan--cross-sectional analysis of the OASIS study. Cerebrovasc Dis. 2010;29(4):361-71. doi: 10.1159/000281834. Epub 2010 Feb 9. PMID 20145390